CLINICAL TRIAL: NCT05663229
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital
Brief Title: Postural Analysis of Patients Receiving Rehabilitation Program
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(II)-20220039
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group-with rehabilitation intervention: We evaluate the static or dynamic posture stability of patients with rehabilitation intervention
  Interventions: Device: Ankle foot orthosis
- Control group-without rehabilitation intervention: We evaluate the static or dynamic posture stability of patients without rehabilitation intervention

INTERVENTIONS:
Device: Ankle foot orthosis — We evaluate the difference of with or without ankle foot orthosis
  Groups: Experimental group-with rehabilitation intervention

SUMMARY:
This is a study for evaluation of posture of patients with neurological disease in rehabilitation department.

DETAILED DESCRIPTION:
In this study, we evaluate the static posture stability of the patient, such as during sitting, standing and dynamic posture stability of the patient, such as during walking, time-up-and-go test.

ELIGIBILITY:
Inclusion Criteria:

* Patient with physical disability followed-up in rehabilitation department

Exclusion Criteria:

* Patients with congitive impairment that can't complete the evalaution well
* Patients with uncontrolled comorbidity diseases
* Attended other study in recent 3 months

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with physical disability followed-up in rehabilitation department
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Displacement of center of gravity during standing | 1 day
  Data collected by motion analysis system
Displacement of center of gravity during walking | 1 day
  Data collected by motion analysis system

SECONDARY OUTCOMES:
Trunk movement | 1 day
  Data collected by motion analysis system
Hip movement | 1 day
  Data collected by motion analysis system
Knee movement | 1 day
  Data collected by motion analysis system
Ankle movement | 1 day
  Data collected by motion analysis system
Foot pressure | 1 day
  Data collected by Pedar (foot pressure system)
Foot reaction force | 1 day
  Data collected by Pedar (foot pressure system) and force plate

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hsuan Tseng, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- aohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No